CLINICAL TRIAL: NCT06012045
Title: A Randomized Controlled Trial of Enhanced Cue Exposure Therapy for Negative Emotional Eating
Brief Title: Enhanced Cue Exposure Therapy for Negative Emotional Eating
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Wai Sze, Principal Investigator, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA220560
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Disordered Eating Behaviors; Binge Eating
Keywords: emotional eating; eating disorders; obesity; exposure and response prevention; behavioral therapy; randomized controlled trial; violation of expectancy; inhibitory learning; habituation; mechanism of change
MeSH Terms: conditions — Disordered Eating Behavior; Bulimia; Emotional Eating; Feeding and Eating Disorders; Obesity; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Cue Exposure Therapy (Experimental): This is the experimental arm. Participants will receive the 6-session enhanced cue exposure therapy.
  Interventions: Behavioral: Enhanced Cue Exposure Therapy
- Behavioral Lifestyle Intervention (Active Comparator): This is the active control arm. Participants will receive the 6-session behavioral lifestyle intervention.
  Interventions: Behavioral: Behavioral Lifestyle Intervention

INTERVENTIONS:
Behavioral: Enhanced Cue Exposure Therapy — The E-CET will consist of six weekly sessions and will be delivered by a clinical psychology trainee in person. Session #1 will be used to introduce to the participant the rationale and procedures of E-CET to establish therapeutic alliance, agreement on treatment goals and tasks, and to collect information on idiosyncratic CS-US expectancies to be targeted in exposures. Sessions #2 to #5 will be in vivo exposures. The interventionist will prompt the participant to evaluate the CS-US expectancy to facilitate the violation of the CS-US expectancy maintaining NEE. Between-session homework exposures will be planned and conducted by the participant in their naturalistic environment. They will also be reviewed at the beginning of the following session to consolidate learning. The final session will consist of consolidation of treatment gains and relapse prevention.
  Arms: Enhanced Cue Exposure Therapy
Behavioral: Behavioral Lifestyle Intervention — The BLI will consist of six weekly sessions of behavioral counselling integrating behavioral strategies for participants to make dietary changes. These behavioral strategies will include education about healthy and balanced diets, goal-setting, problem-solving, and relaxation. A manualized protocol developed by the PI's team for previous studies in the local community will be used.
  Arms: Behavioral Lifestyle Intervention

SUMMARY:
The current study aims to evaluate the efficacy of Enhanced Cue Exposure Therapy (E-CET) in reducing negative emotional eating (NEE), compared to an active control intervention, behavioral lifestyle intervention (BLI), in a parallel-group, participant-blinded, randomized controlled trial. The secondary aim is to evaluate whether changes in conditioned stimulus-unconditioned stimulus (CS-US) expectancies mediate the changes in NEE.

DETAILED DESCRIPTION:
Participants will be randomly assigned to either the experimental treatment or control BLI group. Participants in the experimental group will receive 6 weeks of E-CET treatment and those in the control group will receive 6 weeks of behavioral counselling integrating behavioral strategies for making changes related to diet and exercise. Outcomes will be assessed at baseline, posttreatment, and 3- and 12-month follow-ups.

Research question 1:

Is E-CET an efficacious intervention for reducing NEE?

Hypothesis 1:

E-CET will lead to greater reductions in NEE at posttreatment and follow-up compared to BLI.

Research question 2:

Does E-CET work via the violation of the CS-US expectancies?

Hypothesis 2:

Changes in the believability of CS-US expectancies will mediate the treatment effects of E-CET on NEE.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or over
* a score >3.25 on the emotional eating subscale of the Dutch Eating Behavioural Questionnaire lasting for three months or longer
* confirmed to have, on average, two or more NEE episodes per week using ecological momentary assessments (EMAs)

Exclusion Criteria:

* active suicidal intent or plan
* psychiatric illnesses except mood disorders, anxiety disorders, and eating disorders because mood and anxiety disorders and symptoms are common in those with NEE
* currently receiving psychotherapy, or adjusting to changing psychiatric medication
* substance abuse
* any conditions or circumstances that prevent the participant from receiving all treatment sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Changes in the score on the emotional eating subscale of the Dutch Eating Behaviour Questionnaire (DEBQ) | 14 months (up to 12-month follow-up)
  The subscale consists of 13 items assessing the tendency to eat in response to negative emotions, on a 5-point Likert scale from 1 (never) to 5 (very often). The cutoff point of >3.25 is used to indicate negative emotional eating tendencies. Higher scores indicate greater tendency and severity.
Number of EMA-measured NEE episodes | 14 months (up to 12-month follow-up)
  Participants will respond to fixed-interval prompts asking whether they have engaged in NEE in the assessment period. The sum of all the reported episodes during the seven days will be computed to indicate the frequency of NEE per week.

SECONDARY OUTCOMES:
Changes in NEE | 14 months (up to 12-month follow-up)
  It will be indexed by the association between negative emotionality and caloric consumption measured in three days a week. Negative emotionality will be measured using the four fixed interval prompts per day. Participants will be asked to select the negative emotions applied to them at the moment and rate the intensity of the selected negative emotions on a visual analog scale from 0 (not at all) to 100 (very intense). Caloric consumption will be measured by the 24-hour dietary recall interview conducted for three days a week. Stronger associations will indicate greater NEE.
Changes in caloric consumption | 14 months (up to 12-month follow-up)
  It will be measured by the 24-hour dietary recall interview conducted for three days a week. Nutrition information on food intake (calories, protein, carbohydrates, fat, dietary fibre, sugar, and sodium) will be processed by trained research assistants.
Changes in external eating measured by the external eating subscale of the Dutch Eating Behaviour Questionnaire (DEBQ) | 14 months (up to 12-month follow-up)
  The subscale consists of 10 items assessing the tendency to eat in response to external cues on a 5-point Likert scale from 1 (never) to 5 (very often). Higher scores indicate greater frequencies of disordered eating.
Changes in eating disorder symptoms measured by the Eating Disorder Examination Questionnaire-Short (EDE-QS) | 14 months (up to 12-month follow-up)
  It consists of 12 items assessing the symptoms of eating disorders for the preceding seven days rated on a 4-point Likert scale from 0 (0 days) to 3 (6-7 days). Higher global scores indicate greater eating disorder symptoms.
Changes in body weight | 14 months (up to 12-month follow-up)
  It will be measured in the laboratory using a digital weighing scale.
Changes in mood measured using the Depression, Anxiety and Stress Scale-21 (DASS-21) | 14 months (up to 12-month follow-up)
  The scale consists of 21 items rated on 0 (not at all) to 3 (very much) Likert scales assessing symptoms of anxiety, depression, and stress.
Changes in quality of life measured using the Satisfaction with Life Scale (SWLS) | 14 months (up to 12-month follow-up)
  It is a 5-item scale measuring subjective life satisfaction on a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). Higher total scores indicate greater life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Sze Chan, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data may be shared upon request for research purposes.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified data will become available indefinitely
Access Criteria: Requests to share data will be evaluated by the principal investigator